CLINICAL TRIAL: NCT04707495
Title: Treating Depressed Mood With a Smartphone-delivered Positive Word Stimulation for Subthreshold Depression: Protocol for a Pilot Randomized Controlled Trial
Brief Title: Treating Depressed Mood With a Smartphone-delivered Positive Word Stimulation for Subthreshold Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gunma University (Other)
Responsible Party: Principal Investigator, Kazuki Hirao, Associate Professor, Gunma University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS2020-157
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Subthreshold Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application (SPSRS) (Experimental): The experimental group receives video-viewing intervention using the SPSRS application, which is a smartphone application. SPSRS is programmed to present 150 ms of positive words after presenting 17 ms of self-confidence-boosting words in videos.
  These words are repeated every 5 s. The words to increase self-confidence are "can," "let us try," "good luck," "able," and "do not worry". These self-confidence-boosting words randomly appear in the four corners of the screen. The positive words are "nice," "great," "fantastic," "satisfactory," and "enjoyable". These words are displayed at the center of the screen. Interveners use the SPSRS application according to the operating manual. The participants will use an iPhone managed by interveners to watch a pre-determined 10-minute video.
  Interventions: Device: Smartphone Application (SPSRS)
- Smartphone Application (YouTube) (Active Comparator): The control group uses the same iPhone as the experimental group. The control group uses the YouTube application to receive video-viewing intervention. The control group videos do not show confidence-boosting and positive words. The control group watches the same video as the experimental group for 10 min.
  Interventions: Device: Smartphone Application (YouTube)

INTERVENTIONS:
Device: Smartphone Application (SPSRS) — The experimental group receives video-viewing intervention using the SPSRS application, which is a smartphone application. SPSRS is programmed to present 150 ms of positive words after presenting 17 ms of self-confidence-boosting words in videos.
  These words are repeated every 5 s. The words to increase self-confidence are "can," "let us try," "good luck," "able," and "do not worry". These self-confidence-boosting words randomly appear in the four corners of the screen. The positive words are "nice," "great," "fantastic," "satisfactory," and "enjoyable". These words are displayed at the center of the screen. Interveners use the SPSRS application according to the operating manual. The participants will use an iPhone managed by interveners to watch a pre-determined 10-minute video.
  Arms: Smartphone Application (SPSRS)
Device: Smartphone Application (YouTube) — The control group uses the same iPhone as the experimental group. The control group uses the YouTube application to receive video-viewing intervention. The control group videos do not show confidence-boosting and positive words. The control group watches the same video as the experimental group for 10 min.
  Arms: Smartphone Application (YouTube)

SUMMARY:
Major depressive disorder (MDD) is an important public health problem. Thus, preventive interventions against subthreshold depression (StD), which is one of the key risk factors for the development of MDD, are important. The study developed a smartphone application (SPSRS) that improves depressive symptoms in people with StD by automatically presenting positive word stimuli during videos. The SPSRS application has the potential to improve depressive symptoms in people with StDs. However, whether it can immediately improve depressed moods in people with StD is unclear. The study aims to investigate the immediate effects of SPSRS applications on depressed mood in people with StD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female
2. 20 to 39 years old
3. Beck Depression Inventory-II (BDI-II) score of 10 points or more
4. Persons with written informed consent prior to participation

Exclusion Criteria:

1. History of mental illness
2. Currently receiving treatment from a professional for mental health issues
3. Vision or hearing problems that interfere with daily life.
4. With a major depressive episode in the last two weeks according to the Mini-International Neuropsychiatric Interview

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States 2nd Edition-Adult Short (POMS 2-A Short) | Change of POMS 2-A Short from baseline at the end of 10 minutes of intervention.
  The POMS 2-A Short is a 35-item self-administered questionnaire used to measure mood states. Items are rated using a 5-point Likert-type scale (0 = not at all, 1 = a little, 2 = moderately, 3 = quite a lot, and 4 = extremely). The POMS 2-A Short assesses seven domains, namely, anger-hostility, confusion-bewilderment, depression-dejection, fatigue-inertia, tension-anxiety, vigor-activity, and friendliness. High scores indicate better vigor-activity and friendliness are better but more severe symptoms of the five other domains. In addition, the Total Mood Disturbance (TMD) score is calculated from anger-hostility, confusion-bewilderment, depression-dejection, fatigue-inertia, tension-anxiety, and vigor-activity. TDM is calculated based on a standard value (mean of 50 and standard deviation of 10).

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory State (STAI-S) | Change of STAI-S from baseline at the end of 10 minutes of intervention.
  The STAI is a self-administered questionnaire consisting of two scales that each assesses state anxiety and trait anxiety. Each scale consists of 20 items. Items for STAI-S are scored using a 4-point Likert-type scale (1 = not at all, 2 = somewhat, 3 = moderately so, and 4 = very much so) with the total score ranging from 20 to 80 points. The higher the score, the greater the state anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Gunma University, Maebashi, Gunma, Japan